CLINICAL TRIAL: NCT03499314
Title: A Pilot Trial of Remotely-Supervised Transcranial Direct Current Stimulation (RS-tDCS) to Enhance Motor Learning in Progressive Multiple Sclerosis (MS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-00522
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Multiple Sclerosis
Keywords: Anodal transcranial stimulation (tDCS)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- RS-tDCS Stimulation (Experimental): 20 times 20 minute stimulation session supervised by a study technician through a videoconferencing platform, VSee
  Interventions: Device: Active RS-tDCS +At-Home Manual Dexterity Training; Other: Manual dexterity training
- Sham Stimulation (Placebo Comparator): 20 ×20-minute sessions sham tDCS
  Interventions: Device: Sham RS-tDCS +At-Home Manual Dexterity Training; Other: Manual dexterity training

INTERVENTIONS:
Device: Active RS-tDCS +At-Home Manual Dexterity Training — Bilateral M1-SO electrode placement; Active= anodal 2.0 mA dose × 20 minutes
  Arms: RS-tDCS Stimulation
Device: Sham RS-tDCS +At-Home Manual Dexterity Training — Designed to ensure blinding, includes initial and ending "ramp-up/down" stimulation for 60 seconds
  Arms: Sham Stimulation
Other: Manual dexterity training — Manual dexterity training will be based on the at-home study in MS by Kamm and colleagues, where the training was completed by participants in their homes and demonstrated to be superior to strength training.

SUMMARY:
This is a randomized, double-blind pilot clinical trial to test a novel treatment approach to rehabilitate fine motor function in individuals living with progressive multiple sclerosis (MS) using anodal transcranial direct current stimulation (tDCS) to augment manual dexterity training. Treatment will be delivered to individuals at home using a state-of-the-art remotely supervised tele-rehabilitation protocol, a major advantage for patients with respect to ease of access, feasibility, reinforcement learning and minimal burden of in clinic study visit participation. Improvements in fine motor skill will be assessed at each remote session using a novel portable grip device that measures execution and adaptation or learning of fingertip forces during grasp, which is more sensitive than standard measures of hand function.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS diagnosis, progressive subtype
* 9HPT score between -1.0 and -4.0 standard deviations from age-based normative data
* Score of < 7.5 or less on the EDSS (with caregiver proxy required for those with scores of 6.5 or greater)*
* Ability to understand the informed consent process and provide consent to participate in the study

Exclusion Criteria:

* Primary neurologic, psychiatric or other medical disorder other than MS
* Use of upper extremity Botox injection within 3 months
* Current use of intrathecal Baclofen
* History of seizure disorder
* History of head trauma or medical device in head or neck
* Clinically significant abnormality on EKG
* Symbol Digit Modalities Test or SDMT score ≥3.0 SD from published norms
* WRAT-4 reading level below average (<85) (estimated general intellectual function)
* Skin disorder/sensitive near stimulation locations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RS-tDCS Stimulation | Sham Stimulation
Started | 33 | 32
Completed | 31 | 29
Not Completed | 2 | 3
Not completed — Time Commitment | 1 | 2
Not completed — Medical issue unrelated to research study | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RS-tDCS Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.23 (8.58) | 53.72 (7.62) | 54.49 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 33 | 32 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 28 | 28 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Mean Preload Phase Duration (PLD)
Description: (PLD) is the duration of finger contact until the onset of positive load force. It assesses the time taken to stabilize grasp and is a robust measure of grasp execution.
Time Frame: baseline and 30 minutes for each of 20 sessions, values averaged across sessions
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | RS-tDCS Stimulation | Sham Stimulation
Number analyzed (Participants) | 30 | 24
seconds
  Pre-Stimulation | 0.152 (0.0424) | 0.238 (0.0481)
  Post-Stimulation | 0.163 (0.0426) | 0.202 (0.0476)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | RS-tDCS Stimulation | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 24/33 | 22/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RS-tDCS Stimulation (N=33) | Sham Stimulation (N=32)
Skin Tingling (General disorders) | 17 | 20 — Skin Paresthesia
Skin Itching (General disorders) | 16 | 10 — Skin Paresthesia
Skin Warming (General disorders) | 16 | 7 — Skin Paresthesia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT03499314/Prot_SAP_000.pdf